CLINICAL TRIAL: NCT03062202
Title: The Potential Impact of Using Internet-delivered CBT (iCBT) for People in IAPT Services as a Prequel to High Intensity Therapy (HIT) for Depression and Anxiety Disorders.
Brief Title: Internet-delivered Cognitive Behaviour Therapy at Step 3 of IAPT
Acronym: ICBT@STEP3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derek Richards (Other)
Collaborators: Silver Cloud Health (Other); University of Dublin, Trinity College (Other)
Responsible Party: Sponsor-Investigator, Derek Richards, Director of Clinical Research and Innovation, Silver Cloud Health
Organization: Silver Cloud Health (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICBT@STEP3
Record Dates: First submitted 2017-02-11; First posted 2017-02-23 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Depression; Anxiety
Keywords: Depression; Anxiety; Online interventions; CBT; IAPT
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Depression group (Experimental): SilverCloud iCBT for depression.
  Interventions: Behavioral: SilverCloud
- Anxiety group (Experimental): SilverCloud iCBT anxiety disorders.
  Interventions: Behavioral: SilverCloud
- Comorbid Depression and Anxiety group (Experimental): SilverCloud iCBT for comorbid depression and anxiety.
  Interventions: Behavioral: SilverCloud

INTERVENTIONS:
Behavioral: SilverCloud — SilverCloud Health is a leading provider of online therapeutic solutions to support and promote positive behavior change and mental wellness. SilverCloud delivers interventions for all of the anxiety disorders (panic disorder, social anxiety, phobias, GAD, health anxiety, OCD), depression and also comorbid depression and anxiety. The programs for the treatment of depression and anxiety employ several innovative engagement strategies for improving the user experience. These are divided into several categories: personal, interactive, supportive, and social. Research on the SilverCloud interventions has yielded significant clinical outcomes (Richards et al., 2015).

SUMMARY:
This study will explore the potential impacts of internet-delivered cognitive behavioural therapy (ICBT) at step 3 of the IAPT model. To do this, interventions administered as a prequel to face-to-face therapy will be analysed and compared based on their impacts in regards to access, outcomes (psychological) and costs. A qualitative segment will also be conducted in order to investigate the acceptability and usability of the platform for clinicians and the possibility of developing a therapeutic alliance through an online medium.

DETAILED DESCRIPTION:
Depression and anxiety disorders (panic disorder, social anxiety disorder, specific phobias and generalized anxiety disorder) have been ranked high among the leading causes of disease burden throughout the world, displaying high rates of lifetime incidence, early age onset, high chronicity, and role impairment. Depression and anxiety are associated with impairment in several areas of functioning including social, occupational and personal. The cost to the person and the economy is great, for instance, 105 billion pounds is the estimated cost of depression in the UK with 30% of that being consumed through occupational costs. This has consequently had to be augmented through unemployment benefit to the tune of 7-10 billion.

Improving Access to Psychological Therapies (IAPT):

In 2007 the Department of Health UK announced the introduction of the Improving Access to Psychological Therapies (IAPT) programme. The aim of the programme was to extend access to clinically approved psychological interventions for depression and anxiety. In doing this, the hope was to be able to tackle and help alleviate the burden of psychological distress and its associated costs. In accordance with the model, a five-step approach to psychological care for people with depression and anxiety was introduced and implemented within NHS mental health services The model can be interpreted as a hierarchical care model of mental health, where each step is catered to provide treatment based on the severity of symptoms presented by the patient. This includes watchful waiting by general practitioners care at step 1, step 2 relates to low-intensity psychological interventions, step 3 involves high-intensity psychological interventions, step 4 comprises of specialist mental health care, and step 5 consists of inpatient treatment for mental health problems.

The use of cCBT in IAPT As recommended by the National Institute for Health and Clinical Excellence the IAPT programme offers computerised cognitive behaivoural therapy (cCBT) as a low-intensity, Step 2 intervention for individuals presenting with mild to moderate symptoms of depression and/or anxiety. cCBT and internet-delivered cognitive behavior therapy (iCBT) are delivered by PWPs and support is offered through electronic communication means or by telephone support. However, traditionally they have often suffered with poor engagement and consequently poor clinical outcomes. More recent developments in the field have produced more robust technological platforms, where content is delivered through a variety of media that increase engagement, enhance productivity, and produce better clinical effectiveness. In accordance with what has been utilised in the IAPT model, research has demonstrated the effectiveness of cCBT and iCBT in treating symptoms of depression and anxiety . There is now a substantial body of research evidence that supports the efficacy and effectiveness of online delivered cognitive behavior therapy for depression and anxiety.

Alongside the use of antidepressants, patients at Step 3 IAPT are commonly treated using face-to-face psychological interventions include cognitive behavior therapy, interpersonal therapy, and behavioural activation. In practice, online delivered interventions have been used in some cases for those at step 3 and also as a facilitator for those who are stepping down from Step 3. However, to date, there have not been studies conducted that have examined the potential of online interventions at step 3 and their impact on access rates, clinical and functional outcomes, and costs.

Methodology Objective of the trial To explore the potential of using internet-delivered CBT (iCBT) for people in IAPT services as a prequel to high intensity therapy (HIT) for depression and anxiety disorders.

Research Questions The objective can be further dismantled into;

1. Can SilverCloud achieve positive clinical outcomes for patients?
2. Will patients experience the online intervention as satisfactory?
3. Can an online intervention for depression and anxiety realise cost saving benefits?
4. Do clinicians find the experience of delivering the intervention as satisfactory (usable and acceptable)?
5. Can a therapeutic alliance be established online?

Design The current study will be a mixed methods, uncontrolled feasibility design. The study will utilise both patient and clinician participants. For patients, the study will examine quantitatively clinical outcomes for patients in regards to depression and anxiety, functional outcomes in terms of work and social functioning and cost effectiveness in regards to step-3 services. Therapeutic alliance will also be examined using both patient and clinician participants. Qualitatively, patient satisfaction and clinician experience of the usability and acceptability of the online intervention will be explored. The study will also qualitatively explore the nature of the therapeutic alliance online through use of a semi-structured interview with clinician participants.

ELIGIBILITY:
INCLUSION CRITERIA

* Deemed suitable for an initial Step 3 intervention at IAPT.
* 18 years old and above.
* Able to read English.
* Have capacity to consent.
* Willing to consent.

EXCLUSION CRITERIA

* Flag a risk as per IAPT regulations. (e.g. indicating self-harm on the PHQ-9)
* Receiving an intervention or treatment that is not a part of TAU or another trial.
* Specific communication needs.
* Screened and require an intervention for traumatic stress.
* Do not meet the requirements for step 3 treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2016-12-12; Primary Completion 2017-09-25 (Actual); Study Completion 2017-09-25 (Actual)

PRIMARY OUTCOMES:
Changes in depression symptoms (as measured by the 9 item Patient Health Questionnaire) | Baseline and post-treatment - 8 weeks
  Patient Health Questionnaire-9 (PHQ-9; Kroenke, Spitzer, & Williams, 2001; Spitzer, Kroenke, & Williams, 1999) is a self-report measure of depression that has been widely used in screening, primary care, and research. The PHQ-9 items reflect the diagnostic criteria for depression outlined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition - Text Revision (DSM-IV-TR) (American Psychiatric Association [APA], 2000). Summary scores range from 0-27, where larger scores reflect a greater severity of depressive symptoms. The PHQ-9 has been found to discriminated well between depressed and non-depressed individuals using the clinical cut-off of total score ≥10, with good sensitivity (88.0%), specificity (88.0%) and reliability (.89) (Kroenke et al., 2001; Spitzer et al., 1999).
Changes in anxiety symptoms (as measured by the 7 item Generalised Anxiety Disorder inventory) | Baseline and post-treatment - 8 weeks
  Generalized Anxiety Disorder-7 (GAD-7; Spitzer, Kroenke, Williams, & Löwe, 2006) GAD-7 comprises 7 items measuring symptoms and severity of GAD based on the DSM-IV diagnostic criteria for GAD. The GAD-7 has good internal consistency (α = .92) and good convergent validity with other anxiety scales (Spitzer et al., 2006). Higher scores indicate greater severity of symptoms. The GAD-7 has increasingly been used in large-scale studies as a generic measure of change in anxiety symptomatology, using a cut-off score of 8 (Richards & Suckling, 2009).

SECONDARY OUTCOMES:
Work and Social Adjustment | Baseline and post-treatment - 8 weeks
  Work and Social Adjustment (WASA; Mundt, Marks, Shear & Greist, 2002) is a simple, reliable and valid measure of impaired functioning. It is a simple and reliable (α >.75) 5-item self-report measure which provides an experiential impact of a disorder from the patient's point of view. It looks at how the disorder impairs the patient's ability to function day to day on five dimensions: work, social life, home life, private life and close relationships.
Social Phobia | Baseline and post-treatment - 8 weeks
  Social Phobia Inventory (SPIN, Connor et al., 2000) consists of 17 self-rated items for social anxiety disorder. The test user is required to reflect over the past week and report on their experiences as laid out by the inventory, which assess the domains of social anxiety disorder (fear, avoidance and physiological arousal). Scores are then totaled to produce a value that is representative of symptom severity on a continuum from none to very severe. Internal reliability for the SPIN has been placed at α = .95, with α values for the subscales ranging from .79 - .85.
Obsessive Compulsive Tendencies | Baseline and post-treatment - 8 weeks
  Obsessive-Compulsive Inventory (OCI, Foa et al., 1998) consists of 42 items and 7 subscales, including checking, doubting, washing, ordering, obsessing, hoarding and mental neutralising. Items are presented on a likert scale ranging from 0 (not at all) to 4 (extremely). In total, this scale provides 8 summary scores (7 for the subscales and an overall distress score) and these are represented by mean values. Reliability coefficients for the full scale are placed between .86 - .95 and reliability exceeds .70 for all subscales.
Heath Anxiety | Baseline and post-treatment - 8 weeks
  Short Health Anxiety Inventory (Salkovskis, 2002) measures levels of health anxiety, which is characterized by the misinterpretation of bodily sensations as a serious illness. The shortened version of the scale has been constructed such that it is sensitive to both normal and severe levels of health anxiety. A meta-analysis of the inventory has yielded alpha values between .74 - .96 (Alberts et al., 2013).
Avoidance Behaviours | Baseline and post-treatment - 8 weeks
  Mobility Inventory for Agoraphobia (Chambless et al., 1985) is a scale that was developed in order to measure the avoidance behaviours that are associated with agoraphobia. The α coefficients for both components of the scale are high, with the avoidance alone component yielding α= .96 and avoidance accompanied yielding α = .95 (Chambless et al., 2011)
Responses to Traumatic Events | Baseline and post-treatment - 8 weeks
  Revised Impact of Events Scale (Weiss & Marmar, 1997) is a measure that is typically used with a geriatric population. It looks at typical responses to traumatic events in the domains of intrusion, avoidance, hyperarousal and subjective stress. Full scale reliability analysis yielded α= .96, α= .94 for intrusion, α= .87 for avoidance and α= .91 for hyperarousal (Creamer, Bell & Failla, 2003).
Patient Experience | At the end of the treatment - week 8
  Patient Experience Questionnaire: Will be used to assess patient experience and satisfaction. This questionnaire forms a part of the IAPT minimum data set and is a national requirement in the UK. The PEQ contains several quantitative questions and open ended questions that are used to assess participant's views and satisfaction with service provision.
Therapeutic Alliance for patients | continuous during treatment after each session for 8 weeks
  STAR-P (McGuire-Snieckus, et al., 2007) will be employed to assess patients experience of the therapeutic relationship online. It will be administered post-session.
Usability and Acceptability of the iCBT platforms for clinicians. | At the end of the treatment 2 months
  Usability & Acceptability Questionnaire: At post intervention, the clinicians will be asked to answer open-ended questions regarding their experience that will be administered in an online format. The questions will be formatted into two sections, where the first will consist of items concerning the administration of the programme, and the second will have items examining the process of clinical support online.
Therapeutic Alliance for clinicians | continuous during treatment after each session for 8 weeks
  STAR-C (McGuire-Snieckus, et al., 2007) will be employed to assess clinicians experience of the therapeutic relationship online. The measure will be administered each time the clinician writes a review for their clients.
Qualitative Investigation into Therapeutic Alliance for Clinicians | 1 month post study.
  Semi-structured interview: In addition a sample of clinicians will be invited to take part in a more in-depth interview that will consider key psychological aspect to online delivery of therapy and the nature of the therapeutic relationship online. The interview will be semi-structured and follow a number of key questions that will be developed from the extant literature on therapeutic alliance.

CONTACTS AND LOCATIONS:
Overall Officials: Derek Richards, PhD, Study Director — SilverCloud Health; Jackie Allt, PhD, Principal Investigator — Sussex Community NHS Trust
Locations (1):
- Sussex Community NHS Trust, Brighton, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kessler RC, Berglund P, Demler O, Jin R, Koretz D, Merikangas KR, Rush AJ, Walters EE, Wang PS; National Comorbidity Survey Replication. The epidemiology of major depressive disorder: results from the National Comorbidity Survey Replication (NCS-R). JAMA. 2003 Jun 18;289(23):3095-105. doi: 10.1001/jama.289.23.3095. PMID 12813115
- [Background] Richards D. Prevalence and clinical course of depression: a review. Clin Psychol Rev. 2011 Nov;31(7):1117-25. doi: 10.1016/j.cpr.2011.07.004. Epub 2011 Jul 23. PMID 21820991
- [Background] National Institute for Health and Clinical Excellence. (2006). Computerised cognitive behaviour therapy for depression and anxiety. Technology Appraisal 97. London: National Institute for Health and Clinical Excellence.
- [Background] Gyani A, Shafran R, Layard R, Clark DM. Enhancing recovery rates: lessons from year one of IAPT. Behav Res Ther. 2013 Sep;51(9):597-606. doi: 10.1016/j.brat.2013.06.004. Epub 2013 Jul 4. PMID 23872702
- [Background] Clark DM. Implementing NICE guidelines for the psychological treatment of depression and anxiety disorders: the IAPT experience. Int Rev Psychiatry. 2011 Aug;23(4):318-27. doi: 10.3109/09540261.2011.606803. PMID 22026487
- [Background] National Institute for Clinical Excellence. (2009). The treatment and management of depression in adults (pp. 64). London: UK: National Institute for Clinical Excellence.
- [Background] Layard, R. (2006). The depression report: A new deal for depression and anxiety disorders (No. 15). Centre for Economic Performance, LSE.
- [Background] Cavanagh K, Shapiro DA, Van Den Berg S, Swain S, Barkham M, Proudfoot J. The effectiveness of computerized cognitive behavioural therapy in routine care. Br J Clin Psychol. 2006 Nov;45(Pt 4):499-514. doi: 10.1348/014466505X84782. PMID 17076960
- [Background] Proudfoot J, Ryden C, Everitt B, Shapiro DA, Goldberg D, Mann A, Tylee A, Marks I, Gray JA. Clinical efficacy of computerised cognitive-behavioural therapy for anxiety and depression in primary care: randomised controlled trial. Br J Psychiatry. 2004 Jul;185:46-54. doi: 10.1192/bjp.185.1.46. PMID 15231555
- [Background] Richards D, Richardson T. Computer-based psychological treatments for depression: a systematic review and meta-analysis. Clin Psychol Rev. 2012 Jun;32(4):329-42. doi: 10.1016/j.cpr.2012.02.004. Epub 2012 Feb 28. PMID 22466510
- [Background] Andersson G, Cuijpers P. Internet-based and other computerized psychological treatments for adult depression: a meta-analysis. Cogn Behav Ther. 2009;38(4):196-205. doi: 10.1080/16506070903318960. PMID 20183695
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. Primary Care Evaluation of Mental Disorders. Patient Health Questionnaire. JAMA. 1999 Nov 10;282(18):1737-44. doi: 10.1001/jama.282.18.1737. PMID 10568646
- [Background] American Psychiatric Association (2000). Diagnostic and statistical manual of mental disorders (4th ed., Text Revision). Washington, DC.
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Richards DA, Suckling R. Improving access to psychological therapies: phase IV prospective cohort study. Br J Clin Psychol. 2009 Nov;48(Pt 4):377-96. doi: 10.1348/014466509X405178. Epub 2009 Feb 9. PMID 19208291
- [Background] Mundt JC, Marks IM, Shear MK, Greist JH. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. Br J Psychiatry. 2002 May;180:461-4. doi: 10.1192/bjp.180.5.461. PMID 11983645
- [Background] Connor KM, Davidson JR, Churchill LE, Sherwood A, Foa E, Weisler RH. Psychometric properties of the Social Phobia Inventory (SPIN). New self-rating scale. Br J Psychiatry. 2000 Apr;176:379-86. doi: 10.1192/bjp.176.4.379. PMID 10827888
- [Background] Foa, E. B., Kozak, M. J., Salkovskis, P. M., Coles, M. E., & Amir, N. (1998). The validation of a new obsessive-compulsive disorder scale: The Obsessive-Compulsive Inventory. Psychological Assessment, 10(3), 206.
- [Background] Salkovskis PM, Rimes KA, Warwick HM, Clark DM. The Health Anxiety Inventory: development and validation of scales for the measurement of health anxiety and hypochondriasis. Psychol Med. 2002 Jul;32(5):843-53. doi: 10.1017/s0033291702005822. PMID 12171378
- [Background] Alberts NM, Hadjistavropoulos HD, Jones SL, Sharpe D. The Short Health Anxiety Inventory: a systematic review and meta-analysis. J Anxiety Disord. 2013 Jan;27(1):68-78. doi: 10.1016/j.janxdis.2012.10.009. Epub 2012 Nov 9. PMID 23247202
- [Background] Chambless DL, Caputo GC, Jasin SE, Gracely EJ, Williams C. The Mobility Inventory for Agoraphobia. Behav Res Ther. 1985;23(1):35-44. doi: 10.1016/0005-7967(85)90140-8. No abstract available. PMID 3985915
- [Background] Chambless DL, Sharpless BA, Rodriguez D, McCarthy KS, Milrod BL, Khalsa SR, Barber JP. Psychometric properties of the mobility inventory for agoraphobia: convergent, discriminant, and criterion-related validity. Behav Ther. 2011 Dec;42(4):689-99. doi: 10.1016/j.beth.2011.03.001. Epub 2011 May 24. PMID 22035997
- [Background] Weiss, D. S., & Marmar, C. R. (1997). The impact of event scale-revised. Assessing psychological trauma and PTSD, 2, 168-189.
- [Background] Creamer M, Bell R, Failla S. Psychometric properties of the Impact of Event Scale - Revised. Behav Res Ther. 2003 Dec;41(12):1489-96. doi: 10.1016/j.brat.2003.07.010. PMID 14705607
- [Background] McGuire-Snieckus R, McCabe R, Catty J, Hansson L, Priebe S. A new scale to assess the therapeutic relationship in community mental health care: STAR. Psychol Med. 2007 Jan;37(1):85-95. doi: 10.1017/S0033291706009299. Epub 2006 Nov 9. PMID 17094819
- [Background] Richards D, Timulak L, O'Brien E, Hayes C, Vigano N, Sharry J, Doherty G. A randomized controlled trial of an internet-delivered treatment: Its potential as a low-intensity community intervention for adults with symptoms of depression. Behav Res Ther. 2015 Dec;75:20-31. doi: 10.1016/j.brat.2015.10.005. Epub 2015 Oct 21. PMID 26523885